CLINICAL TRIAL: NCT00441701
Title: Safety and Dose-Ranging Study of the Effects of SCH 527123 in Subjects With Moderate to Severe COPD
Brief Title: Study to Evaluate the Safety and Dose-Range of Navarixin (SCH 527123, MK-7123) in Participants With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) (MK-7123-012)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04592; P04592 (Other: Merck Protocol Number); 2005-004287-23 (EudraCT Number)
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — navarixin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Part 1: Navarixin 3 mg (Experimental): Cohort 1: Participants receive navarixin 3 mg (three 1 mg capsules) once daily (QD) for up to 12 weeks
  Interventions: Drug: Navarixin 1 mg; Drug: Rescue medication
- Part 1: Placebo to navarixin 3 mg (Placebo Comparator): Cohort 1: Participants receive placebo to navarixin (three capsules) QD for up to 12 weeks
  Interventions: Drug: Placebo to match navarixin; Drug: Rescue medication
- Part 1: Navarixin 10 mg (Experimental): Cohort 2: Participants receive navarixin 10 mg (one 10 mg capsule and two placebo capsules) QD for up to 12 weeks
  Interventions: Drug: Navarixin 10 mg; Drug: Placebo to match navarixin; Drug: Rescue medication
- Part 1: Placebo to navarixin 10 mg (Placebo Comparator): Cohort 2: Participants receive placebo to navarixin (three capsules) QD for up to 12 weeks
  Interventions: Drug: Placebo to match navarixin; Drug: Rescue medication
- Part 1: Navarixin 30 mg (Experimental): Cohort 3: Participants receive navarixin 30 mg (three 10 mg capsules) QD for up to 12 weeks
  Interventions: Drug: Navarixin 10 mg; Drug: Rescue medication
- Part 1: Placebo to navarixin 30 mg (Placebo Comparator): Cohort 3: Participants receive placebo to navarixin (three capsules) QD for up to 12 weeks
  Interventions: Drug: Placebo to match navarixin; Drug: Rescue medication
- Part 2: Navarixin 3 mg (Experimental): Cohort 4: Participants receive navarixin 3 mg (three 1 mg capsules) QD for up to 12 weeks
  Interventions: Drug: Navarixin 1 mg; Drug: Rescue medication
- Part 2: Navarixin 10 mg (Experimental): Cohort 4: Participants receive navarixin 10 mg (one 10 mg capsule and two placebo capsules) QD for up to 12 weeks
  Interventions: Drug: Navarixin 10 mg; Drug: Placebo to match navarixin; Drug: Rescue medication
- Part 2: Navarixin 30 mg (Experimental): Cohort 4: Participants receive navarixin 30 mg (three 10 mg capsules) QD for up to 12 weeks
  Interventions: Drug: Navarixin 10 mg; Drug: Rescue medication
- Part 2: Placebo to navarixin (Placebo Comparator): Cohort 4: Participants receive placebo to navarixin (three capsules) QD for up to 12 weeks
  Interventions: Drug: Placebo to match navarixin; Drug: Rescue medication

INTERVENTIONS:
Drug: Navarixin 1 mg — Navarixin 1 mg capsules
  Arms: Part 1: Navarixin 3 mg; Part 2: Navarixin 3 mg
Drug: Navarixin 10 mg — Navarixin 10 mg capsules
  Arms: Part 1: Navarixin 10 mg; Part 1: Navarixin 30 mg; Part 2: Navarixin 10 mg; Part 2: Navarixin 30 mg
Drug: Placebo to match navarixin — Placebo to navarixin capsules
  Arms: Part 1: Navarixin 10 mg; Part 1: Placebo to navarixin 10 mg; Part 1: Placebo to navarixin 3 mg; Part 1: Placebo to navarixin 30 mg; Part 2: Navarixin 10 mg; Part 2: Placebo to navarixin
Drug: Rescue medication — Salbutamol/albuterol - 2 puffs of salbutamol/albuterol approximately every 4 hours as needed for dyspnea relief

SUMMARY:
This is a two-part study conducted at multiple centers, of navarixin (SCH 527123, MK-7123) in participants with moderate to severe chronic obstructive pulmonary disease (COPD). Part 1 of the study is a double-blind, placebo-controlled, randomized, rising-dose study consisting of four treatment groups enrolled in three cohorts. The duration of treatment, for each cohort, will be a 2-week run-in period, followed by a 12-week double-blind treatment period. Treatment initiation for each cohort was staggered by 4 weeks to allow for safety assessment prior to use of higher doses of navarixin. Part 2 of the study will be a double-blind, placebo-controlled, randomized, parallel group study consisting of four treatment groups enrolled as one cohort. The duration of treatment will consist of a 2-week run-in period, followed by a 12-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD based on the American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria.
* >40 to <=75 years of age, of either sex, and of any race.
* Current smoker with at least 10 pack-years of smoking history (eg, 10 pack-year history is equal to smoking 1 pack of cigarettes per day for 10 years or 2 packs per day for 5 years). Participant will be counseled on the risks of smoking and available smoking cessation programs prior to enrollment. Participant who elects to continue to smoke will be eligible for enrollment. Once enrolled, if a participant elects to discontinue smoking, or reduces cigarette consumption, he/she will be allowed to complete the study.
* History of daily sputum production for at least the past 3 months.
* Post-bronchodilator FEV1 must be >=800 mL, and >=40% to <=70% of predicted FEV1.
* Post-bronchodilator ratio of FEV1 to forced vital capacity (FVC) must be <=70%.
* Female participants of childbearing potential must be using a medically acceptable, highly effective, adequate form of birth control (ie, failure rate less than 1% per year when used consistently and correctly) prior to Screening and agree to continue using it while in the study (Screening and Treatment Periods). Medically acceptable, highly effective forms of birth control are hormonal implants, oral contraceptives, medically acceptable prescribed intrauterine devices (IUDs), and monogamous relationship with a male partner who has had a vasectomy.

Female participants should be encouraged to continue using a highly effective method of birth control 30 days following the end of treatment.

* Female participant of child-bearing potential who is not currently sexually active must agree to use a highly effective method of contraception should she become sexually active while participating in the study.
* Male participant must agree to use an adequate form of contraception for the duration of the study and agree to have sexual relations only with women using a highly effective birth control method according to the note for guidance on non-clinical safety studies for the conduct of human clinical trials for pharmaceuticals (CPMP/ICH/286/95 mod).

A highly effective method of birth control is defined as that which results in a low failure rate (ie, less that 1% per year) when used consistently and correctly, such as hormonal implants, injectables, combined oral contraceptives, hormonal IUDs.

* Female participant who is not of childbearing potential must have a medical record of being surgically sterile (eg, hysterectomy, tubal ligation), or be at least 1 year postmenopausal. Absence of menses for at least 1 year will indicate that a female is postmenopausal.
* Capable of complying with the dosing regimen and visit schedules.
* Willing to give written informed consent to participate in the study.

Exclusion Criteria:

* Diagnosed with asthma or other clinically relevant lung disease (other than COPD), eg, sarcoidosis, tuberculosis, pulmonary fibrosis, bronchiectasis, or lung cancer.
* History of previous lung surgery (eg, lobectomy, pneumonectomy, or lung volume reduction).
* Lower respiratory tract infection within 4 weeks prior to the Screening Visit.
* Receiving chronic antibiotic therapy.
* Exacerbation of COPD within the 4 weeks prior to the Screening Visit.
* >20% change at Screening in post-bronchodilator FEV1.
* Female participant who is breast-feeding, pregnant, or intends to become pregnant during the study.
* Clinically relevant medical conditions (eg, hematologic, cardiovascular, renal, hepatic, neurologic, or metabolic).
* Taken inhaled or systemic steroids within 4 weeks of Screening Visit (Visit 1).
* Received an investigational drug within the last 30 days.
* Produced an inadequate amount of sputum at the Screening Visit (Visit 1) or is known to have difficulty producing sputum.
* PBN count of <3000 cells/microliters at Screening Visit (Visit 1).
* Part of the staff personnel directly involved with this study.
* Family member of the investigational study staff.
* Received any study prohibited medication more recently than the indicated washout period, prior to (Screening), or who must continue to receive any prohibited treatment.

Ages: 41 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2006-12-01 (Actual); Primary Completion 2008-10-01 (Actual); Study Completion 2008-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P04592&kw=7123-012&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1: Navarixin 3 mg | Part 1: Placebo to Navarixin 3 mg | Part 1: Navarixin 10 mg | Part 1: Placebo to Navarixin 10 mg | Part 1: Navarixin 30 mg | Part 1: Placebo to Navarixin 30 mg | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Started | 22 | 11 | 22 | 11 | 22 | 11 | 0 | 0 | 0 | 0
Completed | 17 | 7 | 18 | 8 | 20 | 8 | 0 | 0 | 0 | 0
Not Completed | 5 | 4 | 4 | 3 | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Navarixin 3 mg: Cohort 1: Participants receive navarixin 3 mg (three 1 mg capsules) QD for up to 12 weeks
- Total: Total of all reporting groups
Arm/Group | Part 1: Navarixin 3 mg | Part 1: Placebo to Navarixin 3 mg | Part 1: Navarixin 10 mg | Part 1: Placebo to Navarixin 10 mg | Part 1: Navarixin 30 mg | Part 1: Placebo to Navarixin 30 mg | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin | Total
Number analyzed (Participants) | 22 | 11 | 22 | 11 | 22 | 11 | 0 | 0 | 0 | 0 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (5.5) | 57.2 (8.6) | 61.8 (7.3) | 60.2 (7.8) | 56.1 (7.8) | 58.3 (9.4) |  |  |  |  | 57.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 8 | 4 | 8 | 3 |  |  |  |  | 37
  Male | 14 | 5 | 14 | 7 | 14 | 8 |  |  |  |  | 62

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants Who Experience at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, biologic (at any dose), or medical device, which does not necessarily have a causal relationship with the treatment. AEs may include the onset of new illness and the exacerbation of pre-existing conditions. The number of participants who experienced an AE, regardless of causality or severity, was summarized.
Time Frame: Up to 12 weeks
Population: The population consisted of all Part 1 participants who were randomized and received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Part 1: Placebo to Navarixin (Pooled): Pooled Placebo Cohorts: Participants receive placebo to navarixin (three capsules) QD for up to 12 weeks
Arm/Group | Part 1: Navarixin 3 mg | Part 1: Navarixin 10 mg | Part 1: Navarixin 30 mg | Part 1: Placebo to Navarixin (Pooled)
Number analyzed (Participants) | 22 | 22 | 22 | 33
Participants | 10 | 12 | 12 | 20

2. Primary Outcome: Part 1: Number of Participants Who Discontinue Study Drug Due to an AE
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, biologic (at any dose), or medical device, which does not necessarily have a causal relationship with the treatment. AEs may include the onset of new illness and the exacerbation of pre-existing conditions. The number of participants who discontinued study drug, whether permanently or temporarily, due to an AE was summarized.
Time Frame: Up to 12 weeks
Population: The population consisted of all Part 1 participants who were randomized and received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Part 1: Navarixin 3 mg | Part 1: Navarixin 10 mg | Part 1: Navarixin 30 mg | Part 1: Placebo to Navarixin (Pooled)
Number analyzed (Participants) | 22 | 22 | 22 | 33
Participants | 3 | 1 | 2 | 4

3. Primary Outcome: Part 1: Change From Baseline in Absolute Peripheral Blood Neutrophil (PBN) Count
Description: Participants were assessed for absolute PBN counts at Baseline and Week 12. The reported standard deviations (SDs) are pooled across all treatment groups. The rationale for the use of an analysis of variance (ANOVA) method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline and Week 12
Population: The population consisted of all Part 1 participants who were randomized and received at least one dose of study drug and had a Baseline and a Week 12 assessment for absolute PBN count.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part 1: Navarixin 3 mg | Part 1: Navarixin 10 mg | Part 1: Navarixin 30 mg | Part 1: Placebo to Navarixin (Pooled)
Number analyzed (Participants) | 17 | 19 | 20 | 24
10^9 cells/L | -0.33 (1.67) | -1.06 (1.67) | -0.56 (1.67) | 0.06 (1.67)

4. Primary Outcome: Part 2: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1, as measured in liters via spirometry, is a measure of the amount of air expired in 1 second. Participants were to be assessed for pre-bronchodilator FEV1 immediately before dosing with bronchodilator (albuterol sulfate or equivalent) at Baseline and at Week 12. Pre-bronchodilator FEV1 data were to be averaged weekly over the 12-week treatment period for analysis.
Time Frame: Baseline and the Average over 12 weeks
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug, and had a Baseline and at least one post-Baseline assessment for FEV1. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Part 2: Change From Baseline in Daily Morning/Nighttime Sputum Production, Cough, and Dyspnea (SCDS) Score
Description: Participants were to assess their morning (AM) and nighttime (PM) COPD symptoms (sputum production, cough, and dyspnea) on a daily basis in their e-Diaries. Baseline SCDS was defined as the average of AM and PM values over the week prior to and including Day 1 (AM) prior to the first dose of study drug. SCDS data were to be averaged weekly over the 12-week treatment period for analysis.
Time Frame: Baseline and the Average over 12 weeks
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug, and had a Baseline and at least one post-Baseline assessment for AM/PM SCDS scores. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Part 1: Change From Baseline in Percent PBN Count
Description: Participants were to be assessed for percent PBN counts at Baseline and at Week 12.
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 1 participants who were randomized, received at least one dose of study drug, and had a Baseline and a Week 12 assessment for percent PBN count. Since sufficient data for analysis were collected for absolute PBN count, percent PBN count was not assessed.
Arm/Group | Part 1: Navarixin 3 mg | Part 1: Navarixin 10 mg | Part 1: Navarixin 30 mg | Part 1: Placebo to Navarixin (Pooled)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Part 1: Change From Baseline in Sputum Absolute Neutrophil Count (Induced Sputum)
Description: Participants were assessed for induced sputum absolute neutrophil counts via the nebulized method at Baseline and at Week 12. The reported SDs are pooled across all treatment groups. The rationale for the use of an ANOVA method using pooled SD values is the assumption that the SDs are similar across treatment groups.
Time Frame: Baseline and Week 12
Population: The population consisted of all Part 1 participants who were randomized, received at least one dose of study drug, and had a Baseline and Week 12 assessment for induced sputum absolute neutrophil count.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part 1: Navarixin 3 mg | Part 1: Navarixin 10 mg | Part 1: Navarixin 30 mg | Part 1: Placebo to Navarixin (Pooled)
Number analyzed (Participants) | 12 | 18 | 18 | 20
10^9 cells/L | -1.30 (7.83) | -0.84 (7.83) | -4.04 (7.83) | -0.22 (7.83)

8. Secondary Outcome: Part 1: Change From Baseline in Sputum Percent Neutrophil Count (Induced Sputum)
Description: Sputum neutrophils were to be measured as percent of total white blood cells. Participants were to be assessed for induced sputum percent neutrophil counts via the nebulized method at Baseline and at Week 12.
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 1 participants who were randomized, received at least 1 dose of study drug, and had a Baseline and Week 12 assessment for sputum percent neutrophil count. Since sufficient data for analysis were collected for absolute sputum neutrophil count, percent sputum neutrophil count was not assessed.
Arm/Group | Part 1: Navarixin 3 mg | Part 1: Navarixin 10 mg | Part 1: Navarixin 30 mg | Part 1: Placebo to Navarixin (Pooled)
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Part 2: Change From Baseline in Post-Bronchodilator FEV1
Description: FEV1, as measured in liters via spirometry, is a measure of the amount of air expired in 1 second. Participants were to be assessed for post-bronchodilator FEV1 30 minutes after dosing with bronchodilator (albuterol sulfate or equivalent) (reversibility test) at Baseline and Week 12. Post-bronchodilator data were to be averaged weekly over the 12-week treatment period for analysis.
Time Frame: Baseline and the Average over 12 weeks
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug, and had a Baseline and Week 12 efficacy assessment for post-bronchodilator FEV1. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Part 2: Change From Baseline in Forced Expiratory Flow During Middle Half of Forced Vital Capacity (FVC) (FEF25%-75%)
Description: Mid-Breath Forced Expiratory Flow (FEF25%-75%), as measured in liters/minute via spirometry, is the rate at which participants breathe out air from 25 percent of their breath to 75 percent of their breath. Participants were to be assessed for FEF25%-75% at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug, and had a Baseline and Week 12 assessment for FEF25%-75%. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Part 2: Change From Baseline in FVC
Description: FVC, as measured in liters via spirometry, is the amount of air forcibly exhaled from the lungs after taking the deepest breath possible. Post-bronchodilator FVC was to be assessed 30 minutes after bronchodilator administration at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug, and had a Baseline and Week 12 efficacy assessment for FVC. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Part 2: Change From Baseline in Functional Residual Capacity (FRC)
Description: FRC, as measured in liters via body plethysmography, is the volume of air present in the lungs, specifically the parenchyma tissues, at the end of passive expiration. Participants were to be assessed for FRC at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug, and had a Baseline and Week 12 efficacy assessment for FRC. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Part 2: Number of Participants Who Experience a COPD Exacerbation
Description: COPD exacerbation is defined as any change in symptoms or functional status that leads to administration of systemic corticosteroids, antibiotics, an emergency room visit or a hospitalization. The number of participants who experienced a COPD exacerbation was to be summarized.
Time Frame: Up to Week 12
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug, and had a at least one post-Baseline assessment for presence of COPD exacerbation. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Part 2: Change From Baseline in Peak Expiratory Flow (PEF)
Description: PEF, as measured in liters/minute via peak flow meter, is the maximum speed of expiration. Participants were to measure their PEF in triplicate every morning before taking study drug and again every evening.
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug, and had a Baseline and Week 12 efficacy assessment for PEF. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Part 2: Change From Baseline in Induced Sputum Absolute Neutrophil Count
Description: Participants were to be assessed for induced sputum absolute neutrophil counts via the nebulized method at Baseline and at Week 12.
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug and had a Baseline and Week 12 assessment for induced sputum absolute neutrophil count. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Part 2: Change From Baseline in Induced Sputum Percent Neutrophil Count
Description: as for outcome 8
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug and had a Baseline and Week 12 assessment for sputum percent neutrophil count. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Part 2: Change From Baseline in Individual Symptom Scores
Description: Participants were to be assessed for individual symptom scores at Baseline and Week 12 using the following scales: Sputum Production (0=none, unaware of any sputum production to 4=severe, an almost constant problem), Cough (0=none, unaware of coughing to 4=severe, never free of cough or need to cough), and Dyspnea (0=none, unaware of any difficulty to 4=severe, almost constant: present even when resting).
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug and had a Baseline and Week 12 efficacy assessment for individual symptom scores. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Part 2: Change From Baseline in St George's Respiratory Questionnaire (SGRQ) Individual/Total Domains
Description: SGRQ consists of 76 items aggregated into 3 domain scores: Symptoms (frequency/severity), Activity (cause or limited by breathlessness), Impact (social functioning, psychological disturbances from airway disease), and total score. Participants were to assess their symptoms, activity and impact at Baseline and Week 12.
Time Frame: Baseline and Week 12
Population: The population was to consist of all Part 2 participants who were randomized, received at least one dose of study drug and had a Baseline and Week 12 efficacy assessment for SGRQ. Part 2 of this study was not conducted under this protocol.
Arm/Group | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug (Up to 16 weeks)
Description: Part 2 was not conducted under this protocol.
Arm/Group | Part 1: Navarixin 3 mg | Part 1: Navarixin 10 mg | Part 1: Navarixin 30 mg | Part 1: Placebo to Navarixin (Pooled) | Part 2: Navarixin 3 mg | Part 2: Navarixin 10 mg | Part 2: Navarixin 30 mg | Part 2: Placebo to Navarixin
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/22 | 1/22 | 4/33 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 8/22 | 8/22 | 7/22 | 10/33 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Navarixin 3 mg (N=22) | Part 1: Navarixin 10 mg (N=22) | Part 1: Navarixin 30 mg (N=22) | Part 1: Placebo to Navarixin (Pooled) (N=33) | Part 2: Navarixin 3 mg (N=0) | Part 2: Navarixin 10 mg (N=0) | Part 2: Navarixin 30 mg (N=0) | Part 2: Placebo to Navarixin (N=0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Navarixin 3 mg (N=22) | Part 1: Navarixin 10 mg (N=22) | Part 1: Navarixin 30 mg (N=22) | Part 1: Placebo to Navarixin (Pooled) (N=33) | Part 2: Navarixin 3 mg (N=0) | Part 2: Navarixin 10 mg (N=0) | Part 2: Navarixin 30 mg (N=0) | Part 2: Placebo to Navarixin (N=0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 7 (8) | 6 (7) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, eg, any computer access system such as the Internet, World Wide Web, etc.) that report any results of the study.